CLINICAL TRIAL: NCT00272324
Title: Aspirin/Folate Prevention of Large Bowel Polyps
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: 5R01CA059005-12 (NIH)
Record Dates: First submitted 2006-01-03; First posted 2006-01-05 (Estimated); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Colorectal Cancer; Polyps; Adenomas
Keywords: Colorectal neoplasms; Adenomatous polyps
MeSH Terms: conditions — Colorectal Neoplasms; Polyps; Adenoma; Adenomatous Polyps | interventions — Aspirin; Folic Acid

INTERVENTIONS:
Drug: Aspirin
Drug: Folate

SUMMARY:
This is a randomized controlled trial of aspirin and/or folate supplementation for the prevention of the recurrence of neoplastic polyps (adenomas) of the large bowel.

DETAILED DESCRIPTION:
This is a randomized controlled trial of aspirin and/or folate supplementation for the prevention of the recurrence of neoplastic polyps (adenomas) of the large bowel among subjects with a recent history of these tumors. The study is a randomized, double-blind, placebo-controlled trial with a 2 x 3 factorial design.

ELIGIBILITY:
Inclusion Criteria:

1. One neoplastic polyp removed within three months of study entry or within 16 months of study entry if over 1 cm in size or if subject has had a lifetime history of at least two polyps, with the entire large bowel seen by colonoscopy to be free of further polyps within 3 months of entry.
2. An ability and willingness to follow the study protocol, as indicated by the subject's giving informed consent to participate.
3. Good general health, with no severely debilitating diseases or active malignancy that might compromise the patient's ability to complete the study.
4. Anticipated colonoscopic follow-up three years after the qualifying colonoscopy.
5. Age between 21 and 80 years at the time of the intake colonoscopy.
6. For women of childbearing potential, agreement to use effective birth control for the duration of the study.
7. Intent not to take aspirin or aspirin-containing products, NSAIDs or folic acid for the length of the study unless required by a physician.
8. Not randomized previously or currently in a chemoprevention trial, except for the: "Nutritional Prevention of Large Bowel Polyps" Study (Polyps Prevention Study I); and brief participation in the "VA Cooperative Study" with no continuing involvement.

Exclusion Criteria:

1. Invasive carcinoma in any colonic polyp removed.
2. Familial colonic polyposis syndromes.
3. Ulcerative colitis or Crohn's disease.
4. Malabsorption syndrome (e.g. pancreatic insufficiency).
5. Large bowel resection for any reason.
6. Diagnosed narcotic or alcohol dependence
7. Contraindication to aspirin use, including:

   1. documented peptic ulcer disease in the past 20 years
   2. aspirin sensitivity
   3. bleeding diathesis, including hemorrhagic stroke
8. Likelihood of NSAID use

   1. recurring arthritis or other musculo-skeletal problems
   2. frequent NSAID use in 5 years preceding
   3. history of stroke or TIAs
   4. history of angina or myocardial infarction
   5. desire to take aspirin for the prevention of cardiovascular disease
9. Required or contraindicated folic acid use pernicious anemia or folic acid deficiency
10. Pregnancy or lactation.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1121
Dates: Start 1992-02; Study Completion 2007-01

PRIMARY OUTCOMES:
1 or more adenomas | For aspirin: follow-up years 1-3; For folate: follow-up years 1-3 and years 4-8
  colorectal adenomas detected at follow-up colonoscopy

SECONDARY OUTCOMES:
number of adenomas | For aspirin: follow-up years 1-3; For folate: follow-up years 1-3 and years 4-8
  colorectal adenomas detected at follow-up colonoscopy
1 or more advanced lesions | For aspirin: follow-up years 1-3; For folate: follow-up years 1-3 and years 4-8
  adenomas measuring at least 1 cm in diameter or with tubulovillous or villous features, severe dysplasia, or invasive cancer

CONTACTS AND LOCATIONS:
Overall Officials: John A Baron, MD, MSc, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (9):
- United States (8):
  - USC/Kaiser, Los Angeles, California
  - University of Colorado, Denver, Colorado
  - University of Iowa, Iowa City, Iowa
  - Henry Ford Health Sciences Center, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - University of North Carolina, Chapel Hill, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
- University of Toronto, Toronto, Ontario, Canada

REFERENCES:
- [Result] Baron JA, Cole BF, Sandler RS, Haile RW, Ahnen D, Bresalier R, McKeown-Eyssen G, Summers RW, Rothstein R, Burke CA, Snover DC, Church TR, Allen JI, Beach M, Beck GJ, Bond JH, Byers T, Greenberg ER, Mandel JS, Marcon N, Mott LA, Pearson L, Saibil F, van Stolk RU. A randomized trial of aspirin to prevent colorectal adenomas. N Engl J Med. 2003 Mar 6;348(10):891-9. doi: 10.1056/NEJMoa021735. PMID 12621133
- [Derived] Figueiredo JC, Passarelli MN, Wei W, Ahnen DJ, Morris JS, Corley L, Mehta T, Bartley AN, McKeown-Eyssen G, Bresalier RS, Barry EL, Goel A, Hernandez Mesa G, Hamilton SR, Baron JA. Proliferation, apoptosis and their regulatory protein expression in colorectal adenomas and serrated lesions. PLoS One. 2021 Nov 11;16(11):e0258878. doi: 10.1371/journal.pone.0258878. eCollection 2021. PMID 34762658
- [Derived] Passarelli MN, Mott LA, Barry EL, Rees JR, Baron JA. Oral Antibiotics and Risk of New Colorectal Adenomas During Surveillance Follow-up. Cancer Epidemiol Biomarkers Prev. 2021 Oct;30(10):1974-1976. doi: 10.1158/1055-9965.EPI-21-0323. Epub 2021 Jul 21. PMID 34289971
- [Derived] Passarelli MN, Barry EL, Rees JR, Mott LA, Zhang D, Ahnen DJ, Bresalier RS, Haile RW, McKeown-Eyssen G, Snover DC, Cole BF, Baron JA. Folic acid supplementation and risk of colorectal neoplasia during long-term follow-up of a randomized clinical trial. Am J Clin Nutr. 2019 Oct 1;110(4):903-911. doi: 10.1093/ajcn/nqz160. PMID 31401653
- [Derived] Passarelli MN, Barry EL, Rees JR, Mott LA, Ahnen DJ, Baron JA. Body Composition and Aspirin Dose for Colorectal Adenoma Prevention in a Randomized Clinical Trial. Cancer Epidemiol Biomarkers Prev. 2019 Jul;28(7):1262-1265. doi: 10.1158/1055-9965.EPI-19-0205. PMID 31263057
- [Derived] Fedirko V, McKeown-Eyssen G, Serhan CN, Barry EL, Sandler RS, Figueiredo JC, Ahnen DJ, Bresalier RS, Robertson DJ, Anderson CW, Baron JA. Plasma lipoxin A4 and resolvin D1 are not associated with reduced adenoma risk in a randomized trial of aspirin to prevent colon adenomas. Mol Carcinog. 2017 Aug;56(8):1977-1983. doi: 10.1002/mc.22629. Epub 2017 Mar 6. PMID 28218420
- [Derived] Yip WK, Bonetti M, Cole BF, Barcella W, Wang XV, Lazar A, Gelber RD. Subpopulation Treatment Effect Pattern Plot (STEPP) analysis for continuous, binary, and count outcomes. Clin Trials. 2016 Aug;13(4):382-90. doi: 10.1177/1740774516643297. Epub 2016 Apr 19. PMID 27094489
- [Derived] Hazra A, Selhub J, Chao WH, Ueland PM, Hunter DJ, Baron JA. Uracil misincorporation into DNA and folic acid supplementation. Am J Clin Nutr. 2010 Jan;91(1):160-5. doi: 10.3945/ajcn.2009.28527. Epub 2009 Nov 18. PMID 19923375
- [Derived] Cole BF, Baron JA, Sandler RS, Haile RW, Ahnen DJ, Bresalier RS, McKeown-Eyssen G, Summers RW, Rothstein RI, Burke CA, Snover DC, Church TR, Allen JI, Robertson DJ, Beck GJ, Bond JH, Byers T, Mandel JS, Mott LA, Pearson LH, Barry EL, Rees JR, Marcon N, Saibil F, Ueland PM, Greenberg ER; Polyp Prevention Study Group. Folic acid for the prevention of colorectal adenomas: a randomized clinical trial. JAMA. 2007 Jun 6;297(21):2351-9. doi: 10.1001/jama.297.21.2351. PMID 17551129